CLINICAL TRIAL: NCT06439017
Title: Passive Thoughts in Functional Movement Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Aditya Murgai, Passive thoughts in functional movement disorders, Western University, Canada
Other Study IDs: 125294
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-09

CONDITIONS: Functional Movement Disorder
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases with functional movement disorders: The cases will complete the Mind Excessively Wandering Scale (MEWS) and World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0), a 36-item self-administered questionnaire. The individual responses will remain anonymous.
  Interventions: Other: Questionaire
- Healthy controls: The controls will complete the Mind Excessively Wandering Scale (MEWS). The individual responses will remain anonymous.
  Interventions: Other: Questionaire

INTERVENTIONS:
Other: Questionaire — The study will involve completing the Mind Excessively Wandering Scale (MEWS) and World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0), a 36-item self-administered questionnaire.

SUMMARY:
Passive thoughts also known as mind-wandering are the thoughts that are not produced from the current task. When we aren't focused on a task that needs our full attention, our minds tend to drift from one thought to another. It is believed that mind wandering is the baseline or natural state of the mind, and we shift our focus only when needed for a task. Many areas of the brain are active during mind-wandering, and these areas together are called the brain's default network. An important part of this network is the right temporoparietal junction.

Functional movement disorder (FMD) is characterized by unusual movements or walking difficulties that are not caused by a specific brain or nerve injury. Functional movement disorders are believed to be caused due to loss of sense of agency. The sense of agency is the awareness that one is responsible for their own actions. The brain network involved in the sense of agency is mainly located in the right side of the brain, especially in the right temporoparietal junction. In FMD patients, there is decreased connectivity between the right temporoparietal junction and other brain areas that control movement.

Since both passive thoughts (mind wandering) and the sense of agency involve the temporoparietal junction, and because the sense of agency is abnormal in functional movement disorders (FMD), we plan to study passive thoughts in individuals with FMD. The study aims to find out how passive thoughts differ between individuals with FMD and healthy individuals. Passive thoughts will be measured using Mind Excessively Wandering Scale (MEWS).

DETAILED DESCRIPTION:
To evaluate passive thoughts in functional movement disorders (FMD), we will collect data from 30 FMD patients and 30 healthy controls. Patients will be recruited from the movement disorders clinic and the integrated functional movement disorders clinic at LHSC. Both groups will be asked to complete the paper-based Mind Excessively Wandering Scale (MEWS) to evaluate passive thoughts. Additionally, FMD patients will complete the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0), a 36-item self-administered questionnaire designed to measure disability over the past 30 days. Completing both questionnaires will take approximately 15-20 minutes. The questionnaires will be completed once.

ELIGIBILITY:
Inclusion criteria for cases:

1. Diagnosed with a functional movement disorder by the neurologist.
2. Able to understand and read English.

Exclusion criteria for cases:

1. Unable to understand and read English.
2. Diagnosed with dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with a functional movement disorder will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Passive thoughts questionnaire | Day 1
  The Passive Thoughts Questionnaire assesses the severity of passive thoughts and their impact on daily life.

CONTACTS AND LOCATIONS:
Locations (1):
- Aditya Murgai, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No